CLINICAL TRIAL: NCT01758796
Title: A Prospective Randomized Non-inferiority Trial to Compare Operative Versus Non-operative Treatment for ER-stress Positive Weber-B Unimalleolar Fractures
Brief Title: A Noninferiority RCT Comparing Operative vs Nonoperative Treatment for ER-stress Positive Weber-B Unimalleolar Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Harri Pakarinen, Orthopedic surgeon, MD, PhD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OYSrct-Ankle3.2
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Lateral Malleolus Fracture
Keywords: ER-stress positive; Unimalleolar fibula fracture; Operative vs non-operative treatment
MeSH Terms: conditions — Ankle Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Interpretation of data is blinded to treatment group allocation. More precisely, the interpretation of data is carried out without knowledge of the actual treatment given to the particular group, rather labelling groups as "Group 1" and "Group 2". Only then the randomization code is broken, correct data interpretation is chosen, and the draft of the manuscript is finalised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-operative (Experimental): Non-operative treatment with six weeks in a below-the-knee cast. Partial weight-bearing (15 to 20 kilograms) for the first four weeks and then weight-bearing as tolerated for the remaining two weeks.
  Interventions: Procedure: Non-operative treatment
- Surgery (Active Comparator): Open reduction and internal fixation with 1/3 semitubular plate and screws. Post-operatively, surgically treated ankles are placed in a below-the-knee cast for six weeks. They are advised to carry out partial weight-bearing (15 to 20 kilograms) for the first four weeks and then weight-bear as tolerated for the remaining two weeks.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Non-operative treatment — Below-the-knee cast for six weeks.
  Arms: Non-operative
Procedure: Surgery — Open reduction and internal fixation with 1/3 semi-tubular plate and screws.
  Arms: Surgery

SUMMARY:
Current gold standard treatment for unstable (those found unstable in external rotation (ER) stress testing Weber B-type, Lauge-Hansen supination-external rotation type IV) ankle fractures is open reduction and internal fixation (ORIF) with semitubular plates and screws. However, there is some preliminary evidence to suggest that these type of fibula fractures can be managed non-operatively with comparable functional outcome. The aim of this randomized, non-inferiority trial is to assess whether non-operative treatment (cast immobilisation) yields a non-inferior functional outcome compared to surgery with no excess harms (primarily, fracture and wound healing problems and infection).

DETAILED DESCRIPTION:
Seventy per cent of ankle fractures are unimalleolar injuries, the Weber B -type of fibula fracture being by far the most common type. The ankle mortise can either be stable or unstable in this type of fracture depending on the accompanying soft tissue injury. The stability of the ankle mortise has fundamental clinical relevance, as it dictates the subsequent treatment strategy. If left untreated, an unstable ankle mortise may lead to fracture healing complications and increased risk of post-traumatic osteoarthritis and subsequently poor functional outcome. Therefore, current clinical practice guidelines recommend surgical treatment for these injuries. The gold standard surgical treatment for unstable ankle fractures is open reduction and internal fixation (ORIF) using 1/3 semi-tubular plates and screws.

The most common complication following operative treatment of ankle fracture is wound infection, the incidence ranging from 6.1 to10% in unselected patient materials.

To date, there is only one published randomized trial comparing operative and non-operative treatment in patients with an unstable unimalleolar fibula fracture. In this 1-year follow-up, the authors concluded that patients managed nonoperatively had equivalent functional outcomes compared with operative treatment; however, the risk of fracture displacement and problems with union was substantially higher in patients managed nonoperatively. In turn, 10/41 (24%) patients treated operatively were re-operated; five patients had a post-operative infection and five patients required hardware removal.

This prospective randomized non-inferiority trial is designed to compare surgical and non-operative treatment of ER-stress positive unimalleolar ankle fractures. The primary, non-inferiority, intention-to-treat outcome is the Olerud-Molander Ankle Score at 104 weeks or 24 months (OMAS; range, 0-100; higher scores indicating better outcome and fewer symptoms). The predefined non-inferiority margin for the primary outcome at the primary assessment time point is 8 points. Secondary outcomes are ankle function, pain, quality of life, ankle range of motion, and radiographic outcome. Follow-up assessments are performed at 2, 6, 12, and 104 weeks (primary time point). Treatment related complications and harms; symptomatic non-unions, loss of congruity of the ankle joint, and wound infections are also recorded.

The ER-stress test is performed by a consultant trauma orthopedic surgeon or a trauma resident who has completed trauma rotation. Medial clear space opening of 5 mm or more will be considered a positive ER stress test. Patients are randomized to non-operative or surgical treatment using a sealed envelope method. Surgical treatment is carried out using a standard open reduction and internal fixation with 1/3 semitubular plate and screws. Post-operatively, surgically treated ankles are placed in a below-the-knee cast for six weeks. They are advised to carry out partial weight-bearing (15 to 20 kilograms) for the first four weeks and then weight-bear as tolerated for the remaining two weeks. The non-operative treatment protocol is similar to that of the surgically treated patients: six-week below-the-knee cast with partial weight-bearing for the first four weeks and then weight-bearing as tolerated for the remaining two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Weber B unimalleolar ankle fracture
* Age: 16 years or older
* Voluntary
* Operated within 7 days of the trauma
* Walking without aid before accident

Exclusion Criteria:

* Peripheral neuropathy
* Pilon fracture
* Bilateral ankle fracture
* Simultaneous crural fracture
* Pathological fracture
* Active infection around the ankle
* A previous ankle fracture or significant medial ligament trauma
* Lives outside our hospital district or a foreigner
* Co-operation is insufficient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Olerud-Molander Outcome Score (OMAS) | 2 years
  OMAS; scale from 0 to 100, higher scores indicating better outcomes and fewer symptoms. validated, condition-specific, patient-reported measure of ankle fracture symptoms.

SECONDARY OUTCOMES:
The Foot and Ankle Outcome Score (FAOS) | 2 years
  FAOS, 5 subscales from 0-100, with higher scores indicating better function
RAND 36 Health Item Survey (RAND-36) | 2 years
  For health-related quality-of-life. Eight subscales from 0-100, with higher scores indicating better quality of life
a 100 mm Visual Analogue Scale for function and pain (VAS) | 2 years
  Range from 0 to 100, with higher scores indicating more severe pain/dysfunction
Fracture healing | 2 years
  Fracture healing is considered complete when the fracture line disappeared and conversely, those fractures with a visible fracture line are deemed non-unions
Ankle joint movement | 2 years
  Research physiotherapist measures ankle dorsi- and plantarflexion using a goniometer

OTHER OUTCOMES:
Talocrural joint congruence | At two, six and 12 weeks, and at 2 years
  Medial clear space < 4 mm and ≤ 1 mm wider than the superior clear space as measured between the lateral border of the medial malleolus and the medial border of the talus at the level of the talar dome.

CONTACTS AND LOCATIONS:
Overall Officials: Harri J Pakarinen, MD, PhD, Study Director — Oulu University Hospital; Tero HJ Kortekangas, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- OYS, Oulu university hospital, Department of orthopedic and traumatology, Oulu, North Ostrobothnia, Finland

IPD SHARING:
Plan to Share IPD: No
Trial data are not publicly available owing to data privacy, but access to the anonymised dataset can be obtained from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Kortekangas T, Lehtola R, Leskela HV, Taimela S, Ohtonen P, Savola O, Jarvinen TLN, Pakarinen H. Cast immobilisation versus surgery for unstable lateral malleolus fractures (SUPER-FIN): randomised non-inferiority clinical trial. BMJ. 2026 Jan 14;392:e085295. doi: 10.1136/bmj-2025-085295. PMID 41534905

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT01758796/SAP_000.pdf